CLINICAL TRIAL: NCT01779583
Title: Circulating Exosomes As Potential Prognostic And Predictive Biomarkers In Advanced Gastric Cancer Patients: A Prospective Observational Study ("EXO-PPP Study")
Brief Title: Circulating Exosomes As Potential Prognostic And Predictive Biomarkers In Advanced Gastric Cancer Patients ("EXO-PPP Study")
Acronym: EXO-PPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Miguel Servet (Other)
Collaborators: Centro Nacional de Investigaciones Oncologicas CARLOS III (Other); Aragon Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Roberto A. Pazo-Cid, MD, Hospital Miguel Servet
Other Study IDs: EXO-PPP study
Record Dates: First submitted 2013-01-26; First posted 2013-01-30 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Gastric Cancer
Keywords: Advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Serum
  * Tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Advanced gastric cancer patients: Treatment näive advanced gastric cancer patients candidates to first-line chemotherapy
- Control group: Healthy adult volunteers without a cancer diagnosis

SUMMARY:
Exosomes are formed by inward budding of late endosomes, producing multivesicular bodies (MVBs), and are released into the environment by fusion of the MVBs with the plasma membrane. It has been demonstrated that the content and function of exosomes depends on the originating cell and the conditions under which they are produced. Tumor exosome production, transfer and education of bone marrow cells supports tumor growth and metastasis.

In this prospective translational study, preclinical and clinical phases have been designed. On the first step, the main goal is to characterize the molecular profile of gastric cancer derived exosomes. This exosome biosignature may provide a useful diagnostic tool. As a second step, the study will evaluate the prognostic and predictive value of gastric cancer exosomes levels in plasma and kinetics in a prospectively recruited cohort of advanced gastric cancer patients during first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrollment must meet all of the following criteria:

1. Provide signed informed consent. The subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign informed consent, approved by the Independent Ethic Committee (IEC)/Institutional Review Board (IRB) prior to the initiation of any study-specific procedures
2. Men or women aged >= 18 years.
3. Eastern Cooperative Oncology Group Performance Status (ECOG) <= 2.
4. Histologically confirmed adenocarcinoma of the stomach, gastroesophageal junction or esophagus.
5. Metastatic disease or locally advanced disease not amenable to curative surgery.
6. Radiographically assessable, non-measurable disease or measurable disease as per RECIST criteria.
7. Life expectancy of at least 12 weeks from the time of enrollment.
8. No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix.
9. No prior chemotherapy for advanced disease.

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

1. Gastric carcinoid, sarcomas, or squamous cell cancer.
2. Pregnant or lactating females.
3. Significant neurological or psychiatric disorders (psychotic disorders, dementia or seizures) that would prohibit the understanding and giving of informed consent.
4. Active Hepatitis B or C or history of an HIV infection.
5. Active uncontrolled infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be adults with advanced or metastatic gastric cancer (AGC), candidates to receive a first-line systemic therapy, who meet all of the inclusion criteria and none of the exclusion criteria within 28 days prior to the first day of study treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
• Characterization of the molecular profile in tumor derived exosomes from advanced gastric cancer patients undergoing first-line chemotherapy | Up to 2 years from start of study
• Correlation of plasma level and kinetics of gastric cancer derived exosomes (at baseline and monthly during therapy until tumor progression or death) and time-to-event end-points: Overall survival, Progression-free survival and Overall response rate. | Up to 3 years from start of the study

CONTACTS AND LOCATIONS:
Overall Officials: HECTOR PEINADO, PhD, Principal Investigator — Weill Medical College of Cornell University; PILAR MARTIN-DUQUE, PhD, Study Chair — Francisco de Vitoria´s University - Aragon Institute of Health Sciences; ROBERTO A PAZO-CID, MD, Study Director — Aragon Institute of Health Sciences - Medical Oncology Department, Miguel Servet University Hospital
Locations (1):
- Medical oncology Department, Miguel Servet University Hospital, Zaragoza, Spain, Spain

REFERENCES:
- [Background] Peinado H, Aleckovic M, Lavotshkin S, Matei I, Costa-Silva B, Moreno-Bueno G, Hergueta-Redondo M, Williams C, Garcia-Santos G, Ghajar C, Nitadori-Hoshino A, Hoffman C, Badal K, Garcia BA, Callahan MK, Yuan J, Martins VR, Skog J, Kaplan RN, Brady MS, Wolchok JD, Chapman PB, Kang Y, Bromberg J, Lyden D. Melanoma exosomes educate bone marrow progenitor cells toward a pro-metastatic phenotype through MET. Nat Med. 2012 Jun;18(6):883-91. doi: 10.1038/nm.2753. PMID 22635005
- See also: Miguel Servet University Hospital, Zaragoza, Spain — https://maps.google.es/maps?hl=en&q=hospital+miguel+servet+de+zaragoza&bav=on.2,or.r_gc.r_pw.r_cp.r_qf.&bvm=bv.41524429,d.cGE&biw=1067&bih=533&pdl=300&um=1&ie=UTF-8&sa=N&tab=wl
- See also: Francisco de Vitorias´s University (Madrid) — http://www.ufv.es
- See also: Weill Cornell Medical College — http://weill.cornell.edu/